CLINICAL TRIAL: NCT06407180
Title: Efficacy of Intra-Articular Corticosteroid Injections on Clinical Outcomes in Patients With Operative Distal Radius Fractures: A Randomized Controlled Trial
Brief Title: Efficacy of Intra-Articular Corticosteroid Injections on Clinical Outcomes in Patients With Operative Distal Radius Fractures
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Teeradon Waewworawit (Other)
Responsible Party: Sponsor-Investigator, Teeradon Waewworawit, Doctor, Ramathibodi Hospital
Organization: Ramathibodi Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: pending
Record Dates: First submitted 2024-04-30; First posted 2024-05-09 (Actual); Last update posted 2024-05-09 (Actual); Status verified 2024-05

CONDITIONS: Wrist Fractures; Intraarticular Injection
Keywords: Wrist Fractures; intraarticular injection; corticosteroids
MeSH Terms: conditions — Wrist Fractures | interventions — Triamcinolone Acetonide; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intraarticular triamcinolone injection (Experimental): receive Intraarticular triamcinolone injection
  Interventions: Drug: Triamcinolone Acetonide
- placebo group (Placebo Comparator): receive Intraarticular normal saline injection
  Interventions: Drug: Normal saline

INTERVENTIONS:
Drug: Triamcinolone Acetonide — receive intraarticular triamcinolone injection
  Arms: Intraarticular triamcinolone injection
Drug: Normal saline — receive intraarticular normal saline injection
  Arms: placebo group

SUMMARY:
The randomized controlled study which compare clinical outcomes (functional score) in patients with distal radius fractures who underwent open reduction with internal fixation and received intra-articular steroid injections to those who received placebo injections.

DETAILED DESCRIPTION:
Randomization of Patients for Intra-articular Triamcinolone Injection

Objective: To compare the effectiveness of intra-articular Triamcinolone injection versus placebo in patients with distal radius fractures who underwent open reduction with internal fixation

Methods:

Patients: Patients with distal radius fractures who need open reduction with internal fixation procedure Randomization: Patients will be randomly assigned to one of two groups using a block randomization procedure with a block size of 4. Randomization will be performed using STATA version 16.0 software.

Interventions:

Group 1: Patients in this group will receive an intra-articular injection of 10 mg Triamcinolone (1 ml) during surgery.

Group 2: Patients in this group will receive an intra-articular injection of 1 ml normal saline solution during surgery.

Allocation Concealment:

A central randomization service will prepare sealed envelopes containing the assigned treatment for each patient.

The envelopes will be labeled with the patient's name and study ID. The envelopes will be kept in a secure location until the time of surgery.

Blinding:

The study participants, surgeons, and assessors will be blinded to the treatment allocation.

The syringes will be covered with an opaque glove material to further conceal the treatment allocation.

Outcome Measures:

Pain scores Function scores(PRWE score : Patient-Rated Wrist Evaluation) Wrist range of motion Grip strength

Follow-up:

Patients will be followed up at 2 weeks, 6 weeks, 3 months, and 6 months after surgery.

Statistical Analysis:

Demographic Analysis

Analyze the differences in each demographic factor between the groups. For continuous data, use Mean and Standard Deviation (S.D.). For categorical data, use Number, Percentage, and Chi-square. Inferential Statistics

Compare the results of the study, including:

Postoperative pain scores Wrist function score (PRWE) Wrist circumference (mm) Wrist grip strength (kg) Use Mean and S.D. for continuous data. Use Mixed linear model for data analysis. Use STATA 16.0 software for statistical calculations.

ELIGIBILITY:
Inclusion Criteria:

1. Age more than 18 years old
2. Closed unstable distal radius fracture unstable type which need surgical management
3. Received procedure ORIF with plate and screws at injured wrist

Exclusion Criteria:

1. History of corticosteroid allergy
2. Poor Diabetes controlled (HbA1C) > 8
3. Who need Ritonavir while enter this study
4. Unable to follow up until the end of projects
5. Unable to do questionnaires
6. Infection around injured wrist
7. Tear tendon at injured wrist
8. Open fracture of injured wrist

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 58 (Estimated)
Dates: Start 2024-07-01 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Patient-Rated Wrist Evaluation Score | 12 months
  (0-100) Higher scores mean poorer functional outcome

SECONDARY OUTCOMES:
Visual Analog Scale: | 12 months
  (0-10) Higher scores mean more pain
Grip strength (kg) | 12 months
  Measure by hand dynamometer
Wrist circumference | 12 months
ROM of wrist | 12 months
  range of motion

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Mittal A, Bhuti G, Dondeti U, akhtar u, pathak d. CORTICOSTEROID INJECTION AT THE FRACTURE SITE AS AN EFFECTIVE METHOD OF PAIN RELIEF IN SINGLE RIB FRACTURES: A PROSPECTIVE STUDY 2021.
- [Background] Laohaprasitiporn P, Monteerarat Y, Jaderojananont W, Limthongthang R, Vathana T. Validity, Reliability and Responsiveness of the Thai Version of Patient-Rated Wrist Evaluation (Th-PRWE) in Distal Radius Fracture Patients. Siriraj Med J [Internet]. 2021 Mar. 9 [cited 2024 Feb. 15];73(4):275-81. Available from: https://he02.tci-thaijo.org/index.php/sirirajmedj/article/view/246833
- [Result] Court-Brown CM, Caesar B. Epidemiology of adult fractures: A review. Injury. 2006 Aug;37(8):691-7. doi: 10.1016/j.injury.2006.04.130. Epub 2006 Jun 30. PMID 16814787
- [Result] Kong L, Zhai Y, Zhang Z, Lu J, Zhang B, Tian D. Radiocarpal joint stiffness following surgical treatment for distal radius fractures: the incidence and associated factors. J Orthop Surg Res. 2020 Aug 11;15(1):313. doi: 10.1186/s13018-020-01857-6. PMID 32782009
- [Result] Saied A, Heshmati A, Sadeghifar A, Mousavi AA, Arabnejad F, Pooladsanj A. Prophylactic corticosteroid injection in ulnar wrist pain in distal radius fracture. Indian J Orthop. 2015 Jul-Aug;49(4):393-7. doi: 10.4103/0019-5413.159595. PMID 26229158
- [Result] Kim YS, Lee KG, Lee HJ. Effect of triamcinolone acetonide on stiffness after surgical treatment of proximal humerus fractures: a randomized controlled study. Arch Orthop Trauma Surg. 2020 Nov;140(11):1731-1737. doi: 10.1007/s00402-020-03425-3. Epub 2020 Mar 31. PMID 32236715
- [Result] Petersen SK, Hansen I, Andreasen RA. Low frequency of septic arthritis after arthrocentesis and intra-articular glucocorticoid injection. Scand J Rheumatol. 2019 Sep;48(5):393-397. doi: 10.1080/03009742.2019.1584329. Epub 2019 May 31. PMID 31146626
- [Result] Habib GS, Miari W. The effect of intra-articular triamcinolone preparations on blood glucose levels in diabetic patients: a controlled study. J Clin Rheumatol. 2011 Sep;17(6):302-5. doi: 10.1097/RHU.0b013e31822acd7c. PMID 21869712